

IRAS ID: 245270

| Informed Consent Form for Participants | |
|---|---|
| Subject Number: Subject initials: | |
| Title of study: Targeted Metabonomic analysis for Deep Vein Thrombos | sis |
| Please <u>initial</u> the boxes if you agree with the following statements: | |
| I can confirm that I have read and understood the information sheet for this study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. I have received enough information to make up my mind. | |
| I understand that I am free to withdraw from this study, without giving a reason, at any time without my medical care or legal rights being affected. | |
| I agree to: | |
| Disclose my personal medical history to a registered healthcare professional, undertake a physical examination and an ultrasound scan of my legs. | |
| Give blood and urine samples for experimental analysis | |
| For my blood and urine samples and personal identifiable data to be stored securely in Imperial College NHS Trust premises. | |
| For anonymised data relating to my medical history and scan results to be stored in an encrypted file on a secure Imperial College NHS Trust computer. | |
| I give permission for responsible individuals to access my research notes and/or data (i.e. Imperial College, NHS Trust or regulatory authorities) to ensure that the research is being conducted correctly | |
| I give permission for my blood and urine samples to be stored for future use in ethically approved studies (including DNA studies) | |
| I give permission for my registered GP to be informed that I am a participant In this study and of any clinically relevant findings detected during this study | |

| I agree to take part in the above study |
|---|
| Patient SignatureDate |
| (NAME IN CAPITALS) |
| Person taking consent signature |
| (NAME IN CAPITALS) |
| Please tick this box if you would like to be informed of the study results at the end of this research project |